CLINICAL TRIAL: NCT02973750
Title: Determinants of Age-Related Treatment Effectiveness in Ovarian Cancer: Prospective Study of Pharmacokinetics Patterns and Underlying Biology
Brief Title: Determinants of Age-Related Treatment Effectiveness in Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: The V Foundation for Cancer Research (Other); Kay Yow Cancer Fund (Unknown)
Responsible Party: Sponsor
Other Study IDs: MCC-18682
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Ovarian Diseases; Fallopian Tube Diseases; Peritoneal Diseases
Keywords: high-grade serous cancer; stage III cancer; stage IV cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Ovarian Diseases; Fallopian Tube Diseases; Peritoneal Diseases; Neoplasms | interventions — Tissue Banks; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples, Pharmacokinetic (PK) samples, Tumor tissue, Ascites.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pre-Surgery Chemotherapy Patients: All participants. Patients receiving chemotherapy with carboplatin and paclitaxel before their debulking surgery, who may have more chemotherapy after surgery. Sampling procedures will include: Baseline Biopsy; Tissue Collection; Blood Draws.
  Interventions: Procedure: Baseline Biopsy; Procedure: Tissue Collection; Procedure: Blood Draws

INTERVENTIONS:
Procedure: Baseline Biopsy — Baseline biopsy (and ascites fluid sampling if applicable). This is done during the normal work-up procedures.
Procedure: Tissue Collection — Tissue collection during debulking surgery.
Procedure: Blood Draws — Blood samples for paclitaxel and carboplatin plasma levels will be collected in the study. Paclitaxel will be measured on cycle 1 day 1 at predose and then at the end of the infusion, followed by 1, 2, 4, 8 hours after the end of infusion, then on cycle 1 day 2 at 24 hours after the end of infusion. Carboplatin will be sampled for on cycle 1 day 1 at predose and then at the end of the infusion, followed by 0.5, 1.5, 3.5, 7.5 hours after the end of infusion, then on cycle 1 day 2 at 23.5 hours after the end of infusion.

SUMMARY:
While significant progress has been made in the treatment and prognosis of ovarian cancer, this progress has mostly shown benefits for younger women.

This study aims to understand two things: How body composition (the amount of muscle and water versus fat in in the body) affects the dose and side effects of chemotherapy; and the biological reason for the worse prognosis with aging. To get a good view of these effects, investigators are asking the help of both younger and older women for this project.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have one of the following: a) Histological or cytological diagnosis of high-grade serous ovarian, fallopian, or peritoneal cancer, stage III or IV; b) In the opinion of investigator, highly suspicious stage III or IV ovarian, fallopian, or peritoneal cancer (histologically confirmed non-serous ovarian, fallopian, and peritoneal cancers will be considered screening failures).
* At least one biopsiable lesion by CT/US or laparoscopy.
* Have not received previous treatment for ovarian cancer.
* Life expectancy of greater than 6 months.
* Eastern Cooperative Oncology Group (ECOG) performance status <3 (Karnofsky >60%).
* Must have adequate organ and marrow function.
* Deemed eligible for neo-adjuvant chemotherapy with carboplatin and paclitaxel and surgery by their oncologist.
* Women of child-bearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Active second malignancy within last 2 years (except non-melanoma skin cancer or in situ carcinomas.
* Prior treatment for ovarian cancer.
* Potential participants with known brain metastases will be excluded from this clinical trial.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to carboplatin and paclitaxel.
* Known allergy to carboplatin, paclitaxel, or cremophor.
* Uncontrolled concomitant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Women who are pregnant. Breastfeeding should be discontinued if the mother is treated with carboplatin and paclitaxel. These potential risks may also apply to other agents used in this study.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with carboplatin and paclitaxel or other agents administered during the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female cancer patients age 18 years or older, with at least one third of the participants to be aged 70 years or more. Participants must have high-grade serous ovarian, fallopian, or peritoneal cancer, stage III or IV. Women and members of all races and ethnic groups are eligible for this trial. The study is not relevant to men.
  With a sample of 50 patients, investigators can detect a correlation as strong as 0.38 between body composition and AUC of carboplatin and paclitaxel with a power of 0.80 at the significance level of 0.05. In order to allow for a 10% drop out/incompletion rate, investigators will accrue 55 participants.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2020-07-18 (Actual); Study Completion 2020-07-18 (Actual)

PRIMARY OUTCOMES:
Correlation of Skeletal Muscle Index and Fat Index With AUC | 6 months
  Assess the correlation of skeletal muscle index and fat index with the AUC of carboplatin and paclitaxel. Pearson's correlation tests will be performed to assess the correlation of skeletal muscle index and fat index with the AUC of carboplatin and paclitaxel.
Correlation of Skeletal Muscle Index, Fat Index and AUC with Toxicity | 6 months
  Correlate skeletal muscle index, fat index, and AUC with toxicity from preoperative chemotherapy (CTCAE 4.0), nadir neutrophil counts, and relative dose-intensity (RDI). Pearson's correlation tests will be performed to assess skeletal muscle index, fat index, and AUC with toxicity from preoperative chemotherapy, nadir neutrophil counts, and relative dose-intensity (RDI).
Association of Age With Changes | 6 months
  Assess the association of age with changes in mean values, variance, or strength or correlation under 1A and 1B. Unpaired t-tests, Mann-Whitney tests and ANOVA tests will be performed to assess the differences between young (<70) and old (>=70) patients in means, medians and variances of body composition, AUC, toxicity from preoperative chemotherapy, nadir neutrophil counts and RDI.

SECONDARY OUTCOMES:
Correlation of Age With Gene Expression Changes | 6 months
  Assess the correlation with age of gene expression changes in the tumor and its micro-environment before and after neoadjuvant chemotherapy and its correlation with tumor response. Pearson's correlation tests will be performed on age vs. gene expressions, micro-environment and tumor responses before and after neoadjuvant chemotherapy. Paired t-tests will be performed to assess gene expression changes in tumor and its micro-environment before and after neoadjuvant chemotherapy.
Impact of Inflammation on Gene Expression and Response | 6 months
  Assess the impact of inflammation, as assessed by serum and ascites cytokines on gene expression and response, and its correlation with age. Pearson's correlation tests will be performed to assess the impact of inflammation, as assessed by serum and ascites cytokines on gene expression and response, and its correlation with age.
Impact of Inflammation on Toxicity and Relative Dose-Intensity (RDI) | 6 months
  Assess the impact of inflammation on toxicity and RDI. Pearson's correlation tests will be performed to assess the impact of inflammation on toxicity and RDI.

OTHER OUTCOMES:
Relapse Free Survival (RFS) | 12 months
  Correlate the primary and secondary parameters with RFS. Multivariate survival tests using Cox Proportional Hazard model and log-rank tests will be performed to assess the above parameters with relapse-free survival. Given the observational nature of this study, no Bonferroni adjustment is planned.
Overall Survival (OS) | 12 months
  Correlate the primary and secondary parameters with OS. Multivariate survival tests using Cox Proportional Hazard model and log-rank tests will be performed to assess the above parameters with overall survival. Given the observational nature of this study, no Bonferroni adjustment is planned.

CONTACTS AND LOCATIONS:
Overall Officials: Martine Extermann, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/